CLINICAL TRIAL: NCT02126475
Title: L'Expectation Temporelle Dans la Maladie de Parkinson : étude Oculomotrice Psychophysique et Par électroencéphalographie
Brief Title: Temporal Expectations in Parkinson's Disease
Acronym: PEDUPARK
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C12-45; 2012-A01056-37 (Registry Identifier: ID RCB)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Parkinsons Disease; Healthy
Keywords: parkinson patients "ON"; parkinson patients "OFF"; time estimation; anticipation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers
- Park patients

SUMMARY:
Although major progresses were realized during recent years, temporal cognition is still poorly understood. However, abnormal temporal cognition is an underestimated aspect of several neurological disorders, particularly if basal ganglia (BG) are affected. Therefore, the interest of studying temporal cognition is double: firstly, it is an essential function necessary to guide all behavior; secondly, it seems to be very sensitive to the integrity of dopaminergic pathways. It is well known that Parkinson's disease (PD) is partly due to a degeneration of neurons producing dopamine in the Substantia Nigra pars compacta (SNc). Therefore, in this project, PD patients and healthy volunteers will be used as a model to study the role of dopamine in temporal expectation.

An expectation is an internal representation of an event that is likely to occur in the future. Temporal expectation builds-up as time elapses before the upcoming event. The role of temporal expectation in the oculomotor domain has often been studied using anticipatory eye movements as a tool. Indeed, expectation evokes anticipatory eye movements. However, to the knowledge of the investigators, expectation and anticipation have so far been studied in experimental tasks where temporal information is essential but not voluntarily controlled. This is usually referred to as 'automatic' or 'emergent' timing: the timing of the eye movement adapts to the timing of the target, implicitly and without voluntary control of the subject. However, anticipatory movements can also be based on an explicit estimation of time, e.g. during music playing. In summary, timing can be based on cognitive (explicit) or automatic (implicit) processing. The originality of the behavioral task the investigators will use in this study is that it will require an explicit comparison of a memorized duration with elapsing time in order to anticipate target appearance. In this task, expectation of the upcoming event will build up on explicit temporal information.

Same PD patients will be tested under treatment ("ON") and without treatment ("OFF") to determine the effect of dopamine in time expectation . Only levodopa responsive Parkinson patients will be included and among them only those receiving levodopa and/or dopa agonists three times daily at a stable dosis since 30 days.

the investigators hypothesize that eye movements latency will not linearly covary with objective time in "OFF" PD patients. In treated PD patients, a recovery of the linear relationship between subjective and objective time is expected. This would clearly demonstrate the role of dopamine in temporal expectation in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers :

   * Men or women, age: 18 to 65 years old
   * Subject affiliated to a national insurance scheme
   * Informed consent of the study signed
   * Normal neurological exam
2. Patients:

   * Men or women, age: 18 to 65 years old
   * Subject affiliated to a national insurance scheme
   * Informed consent of the study signed
   * Idiopathic Parkinson disease, UKPDSBB criteria (Hughes, Ben-Shlomo, Daniel, & Lees, 1992; Hughes, Daniel, Kilford, & Lees, 1992; Hughes, Daniel, & Lees, 2001)
   * Non fluctuant patients
   * Patients treated by L-Dopa +/- other anti-Parkinsonian's, stable dose for 30 days

Exclusion Criteria:

* Cognitive or behavioural disorder
* Severe psychiatric symptomatology and psychotropic drug use
* Subject non-affiliated to a national insurance scheme
* No signature of the Informed consent of the study
* Subject freedom-deprived by court or administrative order

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and Parkinson patients, non fluctuent
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2016-02-16 (Actual)

PRIMARY OUTCOMES:
oculomotor reaction time: saccade latency | at least 21 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand DEGOS, MD-PhD, Principal Investigator — Département des Maladies du Système Nerveux, Groupe Hospitalier Pitié-Salpêtrière 47-83 boulevard de l'Hôpital 75651 PARIS Cedex 13; Marcus MISSAL, Pr-PhD, Study Director — nstitute of Neurosciences IoNs . Groupe COSY. 53 av. Mounier Boîte B1.53.4 COSY 1200 Bruxelles Belgique; Pierre POUGET, PhD, Study Director — ICM, CNRS, INSERM, Université Pierre et Marie Curie Hôpital de la Salpêtrière 47 boulevard de l'Hôpital 75651 Paris CEDEX 13 France
Locations (2):
- France (2):
  - ICM-IHU, Paris
  - ICM, Paris

REFERENCES:
- [Result] Degos B, Pouget P, Missal M. From anticipation to impulsivity in Parkinson's disease. NPJ Parkinsons Dis. 2022 Oct 3;8(1):125. doi: 10.1038/s41531-022-00393-w. PMID 36184657
- [Result] Degos B, Ameqrane I, Rivaud-Pechoux S, Pouget P, Missal M. Short-term temporal memory in idiopathic and Parkin-associated Parkinson's disease. Sci Rep. 2018 May 16;8(1):7637. doi: 10.1038/s41598-018-25751-8. PMID 29769545